CLINICAL TRIAL: NCT06315361
Title: Prevalence and Clinical Impact of Liver Fibrosis Associated With Non-alcoholic Hepatic Steatosis (NAFLD) in Individuals With Type 2 Diabetes and Relationship With Diabetes Therapies
Brief Title: DIAbetes and NAFLD
Acronym: DIANA
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2445
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: NAFLD; Diabetes; NASH; Fibrosis, Liver; Cirrhosis, Liver; Liver Cancer
Keywords: NAFLD; NASH; Liver fibrosis; Cirrhosis; Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Liver Cirrhosis; Liver Neoplasms; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-alcoholic hepatic steatosis (NAFLD) is characterised by the excessive accumulation of triglycerides in the liver and is often associated, in the absence of significant alcohol consumption, with insulin resistance and metabolic syndrome with which it shares the most frequent clinical manifestations (hypertension, dyslipidaemia, visceral adiposity, glucose intolerance). Due to the pandemic spread of obesity and diabetes and by virtue of better control of viral hepatitis, NAFLD is the most common cause of liver damage in Western countries with a prevalence of around 20-30% of the general population.

The clinical impact of NAFLD in diabetes is considerable and represents a real driver of the major clinical outcomes that impact on the health of the individual, consequently creating a real 'burden of disease' especially in those populations considered to be at higher risk of disease severity.

Individuals with diabetes are, in fact, those at greatest risk of developing the clinical sequelae of NAFLD and often do not receive adequate hepatological support and a correct hepatic pathology. In fact, it has been documented in the literature that the presence of diabetes increases the severity of liver damage, bringing the risk of NASH up to 80% and increasing the risk of significant fibrosis to 30-40% of subjects with hepatic steatosis as well as representing an independent predictor for significant fibrosis. Lastly, the increased risk of hepatocarcinoma in subjects with diabetes and NAFLD should not be overlooked, as documented by our group and confirmed in a large Italian case series.

In subjects with diabetes, moreover, the presence of NAFLD is not only associated with worse glycaemic control, but also with micro- and macro-vascular complications as well as nephrological and neuropathic complications and increased mortality.

Therefore, the possibility of applying the non-invasive fibrosis scores currently available for NAFLD on a large scale, in a population at high risk of progressive liver disease, would make it possible to characterise (a) the true epidemiology of significant fibrosis (F3 or higher); (b) allow primary prevention actions to be carried out by optimising the use of resources or by identifying subjects at greater risk of damage progression; (c) understand, in cases with a long history of disease the true prevalence of clinical outcomes; (d) understand the epidemiology of comorbidities and polypharmacy as a function of significant fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes
* Availability of clinical data for non invasive tests and imaging

Exclusion Criteria:

* Follow-up in clinic at least 1 year

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of significant fibrosis by non invasive tests | 15 years

SECONDARY OUTCOMES:
Identification of MALO (major liver outcomes) | 15 years
Identification of MACE | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Miele, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- UOSD Diabetologia, Catholic University of Rome, Fondazione Policlinico Gemelli IRCCS, Roma, Rome/lazio/italy, Italy